CLINICAL TRIAL: NCT02872649
Title: Pilot-Trial: Dabigatran as an Alternative Anticoagulant in Patients With Left Ventricular Assist Device
Brief Title: Dabigatran as an Alternative Anticoagulant in Patients With Left Ventricular Assist Device (LVAD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: safety reasons
Sponsor: Daniel Zimpfer, MD (Other)
Responsible Party: Sponsor-Investigator, Daniel Zimpfer, MD, MD; Associate Professor of Cardiac Surgery; Principal Investigator, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-024534-38
Record Dates: First submitted 2016-04-02; First posted 2016-08-19 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Thrombosis; Bleeding
MeSH Terms: conditions — Thrombosis; Hemorrhage | interventions — Dabigatran; Phenprocoumon; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- study medication (Experimental): Dabigatran 110mg twice daily with normal renal function (glomerular filtration rate >80 ml/min) Dabigatran 75mg twice daily with impaired renal function (glomerular filtration rate between 80 and 30 ml/min)
  Interventions: Drug: Dabigatran
- control group (Active Comparator): Phenprocoumon dosage according to INR
  Interventions: Drug: Phenprocoumon

INTERVENTIONS:
Drug: Dabigatran
  Other Names: Pradaxa
  Arms: study medication
Drug: Phenprocoumon
  Other Names: Marcoumar; Warfarin
  Arms: control group

SUMMARY:
Patients with severe heart failure supported by left ventricular assist device (LVAD) require adequate long-term anticoagulant therapy. New oral anticoagulants such as the direct thrombin inhibitor dabigatran may represent an alternative to Coumarin for long-term anticoagulation.

In this pilot single-center study, thirty LVAD patients with stable renal function were scheduled to receive phenprocoumon or dabigatran for long-term anticoagulation after implantation of a HeartWare HVAD system following an open-label balanced parallel group design.

ELIGIBILITY:
Inclusion Criteria:

* LVAD (HVAD, Heartware Inc., Framingham, MA, USA) implantation more than one month ago
* Stable renal function (clinical judgement)
* Age 18 years or older
* Ability to give informed consent

Exclusion Criteria:

* Severe chronic renal impairment (CL<30)
* History of significant thromboembolic events
* Significant bleeding disorder
* HIV or Hepatitis C infection
* Heparin induced thrombocytopenia
* Known hypersensitivity to Dabigatran or Phenprocoumon

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-01; Primary Completion 2015-06 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Number of major (life threatening or leading to chronic disability) and minor adverse events due to thromboembolic complications | through study completion, an average of 1 year
Number of major and minor bleeding events (INTERMACS definition) | through study completion, an average of 1 year
  an episode of internal or external bleeding that results in death, the need for re-operation or hospitalization; or necessitates transfusion of red blood cells
Number of patients with necessary treatment changes | through study completion, an average of 1 year
Patient contentment (regular assessment with questionnaire) | Change of Baseline Patient Contentment at 12 months

SECONDARY OUTCOMES:
Treatment effects on INR (coagulation parameter) | 2 weeks, 2 months, 4 months, 6 months, 9 months and 12 months after inclusion
  measured via a blood test
Treatment effects on TT (thrombin clotting time; coagulation parameter) | 2 weeks, 2 months, 4 months, 6 months, 9 months and 12 months after inclusion
  measured via a blood test
Treatment effects on Glomerular Filtration Rate (GFR; renal parameter) | 2 weeks, 2 months, 4 months, 6 months, 9 months and 12 months after inclusion
  measured via a blood test
Treatment effects on Pump Flow (pump parameter), measured in L/min | 2 weeks, 2 months, 4 months, 6 months, 9 months and 12 months after inclusion
Treatment effects on PTT (activated partial thromboplastin time; coagulation parameter) | 2 weeks, 2 months, 4 months, 6 months, 9 months and 12 months after inclusion
  measured via a blood test
Treatment effects on Creatinine (renal parameter) | 2 weeks, 2 months, 4 months, 6 months, 9 months and 12 months after inclusion
  measured via blood test
Treatment effects on Pump Speed (pump parameter), measured in RPM | 2 weeks, 2 months, 4 months, 6 months, 9 months and 12 months after inclusion
Treatment effects on Pump Pulsatility (pump parameter), measured in L/min | 2 weeks, 2 months, 4 months, 6 months, 9 months and 12 months after inclusion
Treatment effects on Pump Power (pump parameter), measured in W | 2 weeks, 2 months, 4 months, 6 months, 9 months and 12 months after inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Univerity Vienna, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andreas M, Moayedifar R, Wieselthaler G, Wolzt M, Riebandt J, Haberl T, Angleitner P, Schloglhofer T, Wiedemann D, Schima H, Laufer G, Zimpfer D. Increased Thromboembolic Events With Dabigatran Compared With Vitamin K Antagonism in Left Ventricular Assist Device Patients: A Randomized Controlled Pilot Trial. Circ Heart Fail. 2017 May;10(5):e003709. doi: 10.1161/CIRCHEARTFAILURE.116.003709. PMID 28500254